CLINICAL TRIAL: NCT04417855
Title: The Effect of Lumbar Disc Herniation on the Kinematics in Lumbo-pelvic Region During Daily Living Activities.
Brief Title: Lumbar Kinematics in People With the Low Back Pain
Status: Completed | Type: Observational
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Tomasz Kuligowski, dr Tomasz Kuligowski, Wroclaw University of Health and Sport Sciences
Other Study IDs: G-Sensor
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Lumbar Disc Herniation; Protrusion; Extrusion of Migrated Disc; Hernia
Keywords: degenerative disc disease; protrusion; extrusion; gait; kinematics
MeSH Terms: conditions — Intervertebral Disc Displacement; Hernia; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LDH: Group of symptomatic individuals with LDH confirmed in MRI.
  Interventions: Diagnostic Test: G-Walk
- Control: Group of asymptomatic individuals with no LDH.
  Interventions: Diagnostic Test: G-Walk

INTERVENTIONS:
Diagnostic Test: G-Walk — Every individual will be examined with a non-invasive "G-Walk" device which is a sensor mounted on a belt and fasten on individuals' lumbar spine region during two test activities: Timed up and go and 6-meter walk tests. Data collection will include kinematic parameters. Oswestry Disability Index (ODI) score will also be collected.

SUMMARY:
This study evaluates the effect of lumbar disc herniation on kinematics in the lumbopelvic region during daily living activities.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is one of the causes of low back pain and contributes to increasing the socio-economic problem. Depending on the reason for the dysfunction, various classifications describing the level of advancement are used. The literature on the subject commonly uses the division into protrusion and extrusion of the intervertebral disc, as approved by the American Society of Neuroradiology.

The lumbopelvic kinematics, including gait and daily living activities, can be affected by the LDH: protrusion or extrusion. This pathology may be different due to the direction of disc migration: centre, left, right or all mentioned. Therefore, we believe that from the different direction of the disc migration the different symptoms can be observed.

ELIGIBILITY:
Inclusion Criteria:

* disc disease located in the lumbar region of the spine confirmed in the MRI
* subacute stage of the disease
* age 18-35 years

Exclusion Criteria:

* advanced degenerative-deformation changes of the spine
* previous fracture of the spine
* neurologic deficits in lower limbs or pelvis
* spondylolisthesis
* transitional vertebra
* rheumatic diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic, students
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test (TUG) | 5 minutes
  The sensor mounted on the belt in lumbar 2nd (L2) vertebra. Following data will be obtained:
  Spatio-temporal parameters standing phase, sitting phase and rotations, trunk kinematics (flexion and/or extension angle) will be collected.
6-meter walking test | 5 minutes
  The sensor mounted on the belt in lumbar 5th (L5) vertebra. Following data will be obtained:
  Total distance travelled general spatio-temporal parameters, variation in spatio-temporal parameters during the 6 minutes walking, pelvis kinematics

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 15 minutes
  The Oswestry Disability Index (ODI) is a valid and reliable assessment tool used by clinicians and researchers to quantify disability for low back pain. The self-completed questionnaire contains ten sections concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.
  For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. After completing, the score is calculated by by summing scores from all sections (total maximum points=50). Total results are calculated as a percentage. The higher the score, the subject's condition is worse.
  The results are interpreted as follows:
  0% to 20%: minimal disability 21%-40%: moderate disability 41%-60%: severe disability 61%-80%: crippled 81%-100%:These patients are either bed-bound or exaggerating their symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- theMedicine, Wroclaw, Lower Silesian Voivodeship, Poland

REFERENCES:
- [Background] Shahvarpour A, Gagnon D, Preuss R, Henry SM, Lariviere C. Trunk postural balance and low back pain: Reliability and relationship with clinical changes following a lumbar stabilization exercise program. Gait Posture. 2018 Mar;61:375-381. doi: 10.1016/j.gaitpost.2018.02.006. Epub 2018 Feb 9. PMID 29448220
- [Background] Kuwahara W, Kurumadani H, Tanaka N, Nakanishi K, Nakamura H, Ishii Y, Ueda A, Deie M, Adachi N, Sunagawa T. Correlation between spinal and pelvic movements during gait and aggravation of low back pain by gait loading in lumbar spinal stenosis patients. J Orthop Sci. 2019 Mar;24(2):207-213. doi: 10.1016/j.jos.2018.09.002. Epub 2018 Oct 12. PMID 30322623
- [Background] Kuai S, Zhou W, Liao Z, Ji R, Guo D, Zhang R, Liu W. Influences of lumbar disc herniation on the kinematics in multi-segmental spine, pelvis, and lower extremities during five activities of daily living. BMC Musculoskelet Disord. 2017 May 25;18(1):216. doi: 10.1186/s12891-017-1572-7. PMID 28545560